CLINICAL TRIAL: NCT04558554
Title: Pharmacy Delivery to Expand the Reach of PrEP in Kenya: Pilot Study
Brief Title: Pharmacy Delivery to Expand the Reach of PrEP in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Katrina Ortblad, Affiliate Assistant Professor, Department of Global Health, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00009587; R34MH120106 (NIH); P30AI027757 (NIH)
Record Dates: First submitted 2020-06-05; First posted 2020-09-22 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: HIV Prevention
Keywords: pre-exposure prophylaxis; Kenya; pharmacy; HIV self-testing; care pathway; pilot

STUDY DESIGN:
Intervention Model Description: During Studies 1a, 1b, and 2, all individuals meeting study and PrEP eligibility criteria will have the option Study 2, study pharmacies will also offer post-exposure prophylaxis (PEP) for HIV prevention to individuals meeting study and PEP eligibility criteria. Also during Study 2, a subset of four study pharmacies (2 per region) will offer STI testing and treatment to individuals meeting study eligibility criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study 1a: Pharmacy-based PrEP delivery Pilot (13 months) (Experimental): Participants in this study will have the option to initiate and/or refill pre-exposure prophylaxis (PrEP) at 4 retail pharmacies in Kenya.
  Interventions: Other: pharmacy-based PrEP delivery
- Study 1b: Pharmacy-based PrEP delivery Refill (12 months) (Experimental): Participants in this study (happening concurrently with Study 1a) will have the option to refill PrEP at 4 retail pharmacies in Kenya after having initiated PrEP at one of 2 public clinics.
  Interventions: Other: pharmacy-based PrEP delivery
- Study 1a: Pharmacy-based PrEP delivery Pilot Extension (6 months) (Experimental): Participants in this study will have the option to initiate and/or refill pre-exposure prophylaxis (PrEP) or initiate PEP at 12 retail pharmacies in Kenya. Additionally, at a subset of 4 pharmacies, participants will have the option to undergo STI testing.
  Interventions: Other: pharmacy-based PrEP delivery

INTERVENTIONS:
Other: pharmacy-based PrEP delivery — The intervention is a new model of PrEP delivery that has never been tried before in an African setting: pharmacy-based PrEP delivery.

SUMMARY:
3 consecutive studies to test a novel model for PrEP initiation and refills in Kenya: pharmacy-based PrEP delivery.

DETAILED DESCRIPTION:
Pre-Exposure Prophylaxis (PrEP) is a new HIV prevention method that works when taken as recommended. To take full advantage of public health benefit of PrEP for HIV prevention, there is need to prioritize access, minimize costs of delivery, and reach out to at-risk populations. In Africa, PrEP is being added to a public health infrastructure which is sometimes burdened by overcrowding and drug stock outs; the ability of health systems to maximize PrEP access necessitates finding novel delivery strategies. Additionally, there exist major barriers to PrEP delivery, which includes stigma, long waiting times, costs of staffing and healthcare providers' unfamiliarity with delivering prevention interventions. In Kenya, and many other resource-limited countries, retail pharmacies (i.e., chemists) fill an important gap in the health care system providing first stop access to treatment, monitoring and preventive care of urgent and prolonged conditions. Potential PrEP users may desire pharmacy-delivered PrEP over facility-delivered PrEP for reasons including increased convenience, increased privacy and greater engagement compared to health facilities that focus on treating ill patients. Retail pharmacies can offer free, subsidized or affordable healthcare services. The core components of PrEP - including HIV testing, adherence and risk reduction counselling, assessment of side effects and provision of refills - are within the scope of practice for pharmaceutical technologists and pharmacists in Kenya. Prior formative qualitative research and a stakeholder meeting led to development of a care pathway for pharmacy-based PrEP delivery (including initiation and refills), endorsed for piloting in a consultation meeting that included a wide spectrum of regulatory, professional, government, and community stakeholders in Kenya. We will conduct 3 separate, consecutive studies.

During Study 1a (13 months), we will pilot this care pathway in 2 retail pharmacies evenly split between 2 different geographies in Kenya: Kisumu and Thika. Activities will include data collection aimed at potential weak points of pharmacy-based PrEP delivery, in domains relating to acceptability, fidelity, and costs.

During Study 1b (12 months, happening concurrently with Study 1a), we will additionally offer pharmacy-based PrEP refills only to clients who initiated PrEP at select public health clinics, to assess how many clients opt to refill PrEP at a study pharmacy (for a fee) as opposed to at the clinic (for free).

During Study 2 (6 months, happening right after Study 1a), we will modify the delivery model (e.g., add new implementation strategies) to address the weak points identified during Study 1a, and we will expand PrEP delivery to six additional retail pharmacies (for a total of 12 pharmacies), evenly split between Kisumu and Thika.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years
* Interested in initiating PrEP at a pilot pharmacy (Study 1a and Study 2), interested in refilling PrEP at a pilot pharmacy (Study 1b), or interested in initiating PEP and/or STI testing at a pilot pharmacy (select pharmacies in Study 2 only)
* Initiated PrEP at a project-affiliated clinic (Study 1b only)
* Meets all criteria (e.g., tests HIV-negative) on checklist for initiating and/or refilling PrEP (all phases), PEP (Study 2 only), and/or STI testing (Study 2 only)
* Able & willing to provide written informed consent

Exclusion Criteria:

* Currently pregnant or breastfeeding (Study 1a & 1b only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1216 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Ortblad, MPH, ScD, Principal Investigator — University of Washington
Locations (2):
- Kenya (2):
  - Kenya Medical Research Institute, Kisumu
  - Kenya Medical Research Institute (Center for Clinical Research - PHRD Thika-Project), Thika

REFERENCES:
- [Derived] Ortblad KF, Kuo AP, Mogere P, Roche SD, Kiptinness C, Wairimu N, Gakuo S, Baeten JM, Ngure K. Low selection of HIV PrEP refills at private pharmacies among clients who initiated PrEP at public clinics: findings from a mixed-methods study in Kenya. BMC Health Serv Res. 2024 May 11;24(1):618. doi: 10.1186/s12913-024-10995-0. PMID 38730398
- [Derived] Ortblad KF, Mogere P, Omollo V, Kuo AP, Asewe M, Gakuo S, Roche S, Mugambi M, Mugambi ML, Stergachis A, Odoyo J, Bukusi EA, Ngure K, Baeten JM. Stand-alone model for delivery of oral HIV pre-exposure prophylaxis in Kenya: a single-arm, prospective pilot evaluation. J Int AIDS Soc. 2023 Jun;26(6):e26131. doi: 10.1002/jia2.26131. PMID 37306128
- [Derived] Omollo V, Asewe M, Mogere P, Maina G, Kuo AP, Odoyo J, Oware K, Baeten JM, Kohler P, Owens T, Bukusi EA, Ngure K, Ortblad KF. The Fidelity of a Pharmacy-Based Oral HIV Pre-Exposure Prophylaxis Delivery Model in Kenya. J Acquir Immune Defic Syndr. 2023 Aug 15;93(5):379-386. doi: 10.1097/QAI.0000000000003208. PMID 37079900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pharmacists recruited participants by hanging up promotional posters encouraging clients to ask about PrEP (or PEP, in Study 2 only) for HIV prevention. They also offered to screen clients who were purchasing products indicative of sexual activity and potential HIV exposure (e.g., emergency contraception, pregnancy testing, STI treatment). Participants in Study 1a & b were recruited from Nov.2020-Dec. 2021 and in Study 2 from Jan.-Jul. 2022.
Groups:
- Study 1a: Pharmacy-based PrEP Delivery Pilot (13 Months): Participants in this study will have the option to initiate and/or refill pre-exposure prophylaxis (PrEP) at 4 retail pharmacies.
- Study 1b: Pharmacy-based PrEP Refill (12 Months): Participants in this study (happening concurrently with Study 1a) will have the option to refill PrEP at 4 retail pharmacies after having initiated PrEP at one of 2 public clinics.
- Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months): Participants in this study will have the option to initiate and/or refill pre-exposure prophylaxis (PrEP) or initiate PEP at 12 retail pharmacies. Additionally, at a subset of 4 pharmacies, participants will have the option to undergo STI testing.
Period: Overall Study
Arm/Group | Study 1a: Pharmacy-based PrEP Delivery Pilot (13 Months) | Study 1b: Pharmacy-based PrEP Refill (12 Months) | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Started | 287 | 106 | 823
Completed | 287 | 106 | 823
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cumulative number of participants who, across Study 1a, 1b, and 2, consented and initiated PrEP or PEP at a study pharmacy.
Groups:
- Study 1b: Pharmacy-based PrEP Delivery Refill (12 Months): Participants in this study (happening concurrently with Study 1a) will have the option to refill PrEP at 4 retail pharmacies after having initiated PrEP at one of 2 public clinics in Kenya.
- Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months): Participants in this study will have the option to initiate and/or refill pre-exposure prophylaxis (PrEP) or initiate PEP at 12 retail pharmacies in Kenya. Additionally, at a subset of 4 pharmacies, participants will have the option to undergo STI testing.
- Total: Total of all reporting groups
Arm/Group | Study 1a: Pharmacy-based PrEP Delivery Pilot (13 Months) | Study 1b: Pharmacy-based PrEP Delivery Refill (12 Months) | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months) | Total
Number analyzed (Participants) | 287 | 106 | 823 | 1216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 287 | 106 | 823 | 1216
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [22 to 33] | 31 [26 to 38] | 25 [22 to 31] | 26 [22 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 63 | 429 | 616
  Male | 163 | 43 | 394 | 600
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 287 | 106 | 823 | 1216

OUTCOME MEASURES:

1. Primary Outcome: PrEP Initiation
Description: Cumulative number of participants who initiated PrEP at pilot pharmacies (during Study 1a and Study 2) among those eligible for pharmacy PrEP services.
Time Frame: Over 13-month duration of Study 1a and 6-month duration of Study 2
Population: Participants eligible for pharmacy PrEP among those screened. PLEASE NOTE: Prospective study participants were screened for preliminary eligibility for PrEP before they were enrolled in the study. Across Study 1a and 2, 1603 clients were screened and found eligible for PrEP; however, not all of these clients decided to enroll in the study. That is why this number exceeds the number who started the study (n=1216) reported in other sections of this record.
Measure: Count of Participants; unit: Participants
Groups:
- Study 1a: Pharmacy-based PrEP Delivery Pilot (13 Months): During Phases 1a and 2, participants in this experimental arm (which includes all participants) will have the option to initiate and/or refill pre-exposure prophylaxis (PrEP) at retail pharmacies in Kenya.
Arm/Group | Study 1a: Pharmacy-based PrEP Delivery Pilot (13 Months) | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 575 | 1028
Participants | 287 | 661

2. Primary Outcome: PrEP Retention
Description: For Study 1a and 2: Percentage of participants who refilled PrEP at a pilot pharmacy, among those who initiated PrEP at a pilot pharmacy.
  Study 1b: Percentage of participants who refilled PrEP either at a pilot pharmacy or at a pilot clinic, among those who initiated PrEP at a pilot clinic.
Time Frame: Over 13-month duration of Study 1a, 12-month duration of Study 1b, and 6-month duration of Study 2
Population: For Study 1a and 2: Number of participants who initiated PrEP at a pilot pharmacy.
  Study 1b: Number of participants who initiated PrEP at a pilot clinic. PLEASE NOTE: This denominator (n=1054) exceeds the number of clients reported as having initiated PrEP for our primary outcome measure of "PrEP initiation" (n=948) because it includes 106 clients who, as part of Study 1b, had initiated PrEP at a pilot clinic.
Measure: Count of Participants; unit: Participants
Groups:
- Study 1a: Pharmacy-based PrEP Delivery (13 Months): Participants in this study will have the option to initiate and/or refill pre-exposure prophylaxis (PrEP) at 4 retail pharmacies in Kenya.
- Study 1b: Pharmacy-based PrEP Refill (12 Months): Participants in this study (happening concurrently with Study 1a) will have the option to refill PrEP at 4 retail pharmacies in Kenya after having initiated PrEP at one of 2 public clinics.
Arm/Group | Study 1a: Pharmacy-based PrEP Delivery (13 Months) | Study 1b: Pharmacy-based PrEP Refill (12 Months) | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 287 | 106 | 661
Participants
  Any PrEP continuation | 153 | 41 | 476
  No PrEP continuation | 134 | 65 | 185

3. Secondary Outcome: PEP Initiation
Description: Study 2: Number of participants who initiated PEP at a pilot pharmacy.
Time Frame: Over 6-month duration of Study 2
Population: Study 2: Number of participants who were screened and found preliminarily eligible for PEP.
Measure: Count of Participants; unit: Participants
Groups:
- Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months): During Study 2, participants will also have the option to initiate post-exposure prophylaxis (PEP) at a study pharmacy.
Arm/Group | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 192
Participants | 162

4. Secondary Outcome: Selection of Pharmacy-based PrEP Refills
Description: Study 1b: Percentage of participants who initiated PrEP at a clinic and subsequently opted to refill their PrEP prescription at a pilot pharmacy.
Time Frame: During the 12-month duration of Study 1b
Population: Study 1b: Number of participants who initiated PrEP at a pilot clinic and were given the option to refill at a pilot pharmacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 1b: Pharmacy-based PrEP Delivery Refill (12 Months)
Number analyzed (Participants) | 106
Participants | 3

5. Secondary Outcome: PrEP Adherence
Description: Study 1a and Study 2: Percentage of randomly selected DBS samples with drug concentrations indicating PrEP adherence
Time Frame: Over 12-month duration of Study 1a and the 6-month duration of Study 2
Population: Study 1a and Study 2: Number of DBS samples randomly selected for drug concentration testing. Note: DBS samples were only collected from participants who had initiated PrEP at a pilot pharmacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 1a: Pharmacy-based PrEP Delivery (13 Months) | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 61 | 48
Participants | 16 | 16

6. Secondary Outcome: STI Testing Uptake
Description: Study 2: Number of participants who opt to undergo STI testing (provide a urine sample for lab-based testing) at pilot pharmacies
Time Frame: Over 6-month duration of Study 2
Population: Study 2: Number of participants who were screened and found potentially eligible for STI testing (providing a urine sample for lab-based testing) at pilot pharmacies. NOTE: STI testing was only offered at a sub-section of study pharmacies (n=4)
Measure: Count of Participants; unit: Participants
Arm/Group | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 64
Participants | 53

7. Secondary Outcome: Transition From PEP to PrEP
Description: Study 2: Percentage of participants who completed the full PEP regimen and subsequently initiated PrEP at a pilot pharmacy, among those who initiated PEP at a pilot pharmacy,
Time Frame: Over 6-month duration of Study 2
Population: Study 2: Number of participants who initiated and completed PEP regimen at a pilot pharmacy
Measure: Count of Participants; unit: Participants
Arm/Group | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 162
Participants | 30

8. Secondary Outcome: PrEP Initiation Among STI Testing Clients
Description: Study 2: Number of participants who come to a study pharmacy for STI testing, undergo STI testing, and initiate PrEP at the pilot pharmacy during the same study visit or a subsequent study visit
Time Frame: Over 6-month duration of Study 2
Population: Phase 2: Number of participants who underwent STI testing at a pilot pharmacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 53
Participants | 45

9. Secondary Outcome: Selection of Option to Self-administer HIV Risk Assessment Screening Tool
Description: Study 2: Number of participants who opt to self-administer the HIV Risk Assessment Screening Tool (as opposed to having the pharmacy provider administer it)
Time Frame: Over 6-month duration of Study 2
Population: Phase 2: Number of participants who completed screening for PrEP/PEP eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
Number analyzed (Participants) | 823
Participants | 151

ADVERSE EVENTS:
Time Frame: Phase 1a: 13 months Phase 1b (concurrent with Phase 1a): 12 months Phase 2: 6 months Total duration from start of Phase 1a (Nov. 2020) to completion of Phase 2 (July 2022): 20 months
Arm/Group | Study 1a: Pharmacy-based PrEP Delivery Pilot (13 Months) | Study 1b: Pharmacy-based PrEP Refill (12 Months) | Study 2: Pharmacy-based PrEP Delivery Pilot Extension (6 Months)
All-Cause Mortality (participants affected / at risk) | 0/287 | 0/106 | 0/823
Serious Adverse Events (participants affected / at risk) | 0/287 | 0/106 | 0/823
Other Adverse Events (participants affected / at risk) | 0/287 | 0/106 | 0/823

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04558554/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04558554/SAP_001.pdf
  • Informed Consent Form (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04558554/ICF_002.pdf